CLINICAL TRIAL: NCT01678118
Title: Tobacco-Focused Patient Navigation to Address Barriers to Utilization of Community-Based Smoking Cessation Services in Primary Care
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sophie Davis School of Biomedical Education at The City College of New York (Unknown); NYU Langone Health (Other); Ralph Lauren Center for Cancer Care and Prevention (Other); Heritage Health Center, New York (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11-028
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Minority Smokers
Keywords: Patient Navigation; Tobacco dependent; smoking; Cessation; 11-028
MeSH Terms: conditions — Smoking | interventions — Patient Navigation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- minority smokers: A single arm ABA design will be used to pilot a tobacco-focused patient navigation (TPN) intervention for low income, minority smokers.
  Interventions: Behavioral: Patient Navigator

INTERVENTIONS:
Behavioral: Patient Navigator — The pt navigator will phone (email, text, or other preferred method of contact) pts prior to the date of previously set individual goals (e.g. going to an appt, getting their cessation medications filled, etc) as a reminder & to discuss barriers such as finances, transportation or ambivalent motivation. In this manner, pts receive navigation services tailored to their individual needs & barriers. Once pts are connected with a cessation service (defined as either using cessation medication or at least 1 contact with a Quitline or community-based cessation counselor)or provider-prescribed cessation medication usage, continues the navigation intervention will be considered complete. W/I the 3 month engagement period, pts will receive up to 6 contacts from the Pt Navigator following referral from primary care provider. Consistent with recommended pt navigation practice, the navigator will provide feedback to primary care provider regarding cessation services that the pts are receiving.

SUMMARY:
Patient navigators have been shown to assist people seeking cancer screening and other medical services. The purpose of this study is to see whether a patient navigator can link smokers to available community resources shown to help smokers quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Self-reported current daily smoker, as verified with a portable alveolar carbon monoxide (CO) analyzer (24 hour point prevalence); CO levels ≥ 8 ppm.
* English and/or Spanish-speaking
* Referred to the navigation program by their primary care clinician
* At baseline, participants report at least thinking about quitting (i.e., Contemplation or Preparation stages of readiness to quit).

Exclusion Criteria:

* Serious, untreated psychiatric illness (e.g., schizophrenia,) or active substance abuse likely to preclude adherence to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will also be recruited from Heritage Health Center, located at 1727 Amsterdam Ave, which serves a large proportion to low income, minority patients in Harlem, New York. Also, from the Ralph Lauren Center for Cancer Care and Cancer Prevention (RLCCCP), a community based Center for the prevention, diagnosis, and treatment of cancer located at 1919 Madison Avenue.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
patient navigation (TPN) feasibility | 1 year
  To evaluate the study's potential in terms of its reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) of the intervention, tobacco-dependent patients will be asked to complete an intake interview and a telephone follow-up interview (at 3 to 6 months post-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Heritage Health Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/